CLINICAL TRIAL: NCT04842903
Title: Effect of Therapeutic Touch on Sleep Quality and Anxiety in Individuals With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial
Brief Title: Effect of Therapeutic Touch on Sleep Quality and Anxiety in Individuals With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Çalışkan, Research Assisstant, Abant Izzet Baysal University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-SBF-MAC-01
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: COPD; Anxiety; Sleep
Keywords: Chronic obstructive pulmonary disease; Therapeutic touch; Sleep quality; Anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Therapeutic touch and standard nursing care of the clinic (such as breathing exercise, postural drainage) was applied.
  Interventions: Other: Therapeutic Touch
- Control Group (No Intervention): Only standard nursing care of the clinic (such as breathing exercise, postural drainage) was applied.

INTERVENTIONS:
Other: Therapeutic Touch — Therapeutic touch is an energy transfer process based on the assumption that every living organism in the universe has an energy field and these energy fields that interact with each other can be changed with the practices made by a conscious and certain intent. TT is an independent nursing practice first applied and developed by nurses Dora Kunz and Dolores Krieger in 1972. TT is also an art of concentration therapy in which the therapist focuses on consciousness as a focus to create balance and coordination in the mutual energy fields of the patient and the environment, and uses their hands to transfer energy. The fact that TT is easy to use, has no known side effects, has low costs, is non-invasive, and its importance among nurses and increasing frequency of its practice in recent years show that it is a powerful alternative to other CAT methods.
  Arms: Experimental Group

SUMMARY:
Purpose: The purpose is to determine the effect of therapeutic touch on the sleep quality and anxiety of individuals with chronic obstructive pulmonary disease.

Material and methods: This study was conducted between March 2018 and March 2019 as a randomized controlled experimental study conducted with pre-test post-test model. In addition to the routine nursing care, therapeutic touch (TT) and study scales were applied to the experimental group for a total of three sessions, once a day and 10 minutes each, for three consecutive days and only study scales were applied to the control group. The data was collected using Personal Information Form, Richard-Campbell Sleep Questionnaire and State Anxiety Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Literate
* Oriented, open to communication and cooperation
* Those who are hospitalized in the clinic for at least four days
* Patients who volunteered to participate in the study were included.

Exclusion Criteria:

* Have any diagnosed psychiatric disorder
* Using antidepressants, antihistamines, benzodiazepines, hypnotic and narcotic drugs
* Persons using any other complementary and alternative treatment method during the therapeutic touch application were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Richard-Campbell Sleep Questionnaire | 3 days
  It was developed by Richards in 1987. It is a five-item scale that evaluates depth of night sleep, duration of falling asleep, frequency of awakening, duration of being awake when waking up and sleep quality. Each item in the scale is evaluated on a chart between 0 and 100 with visual analogue scale. The minimum score that can be obtained from the scale is 100, and the minimum score is 0. The higher the score on the scale, the higher the sleep quality. The Cronbach alpha coefficient of the scale, developed by Richards was 0.82.

SECONDARY OUTCOMES:
State Anxiety Inventory | 3 days
  It was developed by Spielberger et al in 1970. State anxiety inventory measures the anxiety levels of individuals aged 14 years. The scale consists of 20 items. In the scale, participants are asked to mark one of the options "never = 1", "a little = 2", "a lot = 3", "totally = 4" according to the severity of the emotions, thoughts or behaviors they express. The highest score that can be obtained from the scale is 80 and the lowest score is 20. The higher the total scale score, the higher the anxiety level of the individual filling the scale. Spielberger et al. Stated that 0-19 points obtained from the scale are not anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-80 points mean severe anxiety, individuals with a score of 60 and above need professional help.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül CERİT, PhD, Study Director — Bolu Abant Izzet Baysal University Faculty of Health Science
Locations (1):
- Bolu Abant Izzet Baysal Univercity, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caliskan MA, Cerit B. Effect of therapeutic touch on sleep quality and anxiety in individuals with chronic obstructive pulmonary disease: A randomized controlled trial. Complement Ther Clin Pract. 2021 Nov;45:101481. doi: 10.1016/j.ctcp.2021.101481. Epub 2021 Sep 8. PMID 34536666